CLINICAL TRIAL: NCT03636165
Title: Pre-emptive Scalp Infiltration With Ropivacaine Plus Methylprednisolone vs Ropivacaine Alone for Relief of Postoperative Pain After Craniotomy in Children (RP/MP vs RP)
Brief Title: Scalp Infiltration With Methylprednisolone Plus Ropivacaine for Post-Craniotomy Pain in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY 2018-066-02-1
Record Dates: First submitted 2018-08-02; First posted 2018-08-17 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Pain, Postoperative; Post-Craniotomy Headache
Keywords: Postoperative Pain; Post-Craniotomy Headache; Methylprednisolone; Ropivacaine; Pre-emptive Scalp Infiltration; Child
MeSH Terms: conditions — Pain, Postoperative | interventions — Methylprednisolone; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MP plus RP group (Experimental): Patients in RP/MP group will receive a peri-incisional scalp infiltration with 0.125% methylprednisolone and 0.2% ropivacaine and normal saline miscible liquids. The assigned solution will be injected subcutaneously by surgeons along the incision and throughout the entire thickness of the scalp before skin incision. The volume of local infiltration solution will be decided by surgeons according to the cut length, and the capacity of the solution will be recorded by investigators.
  Interventions: Drug: Methylprednisolone; Drug: Ropivacaine
- RP group (Active Comparator): Patients in RP group will receive peri-incisional scalp infiltration with 0.2% ropivacaine alone. The assigned solution will be injected subcutaneously by surgeons along the incision and throughout the entire thickness of the scalp before skin incision. The volume of local infiltration solution will be decided by surgeons according to the cut length, and the capacity of the solution will be recorded by investigators.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Methylprednisolone — The local infiltration solution containing 1.25mg Methylprednisolone per milliliter.
  Arms: MP plus RP group
Drug: Ropivacaine — The local infiltration solution containing 2mg Ropivacaine per milliliter.

SUMMARY:
At present, pediatric postoperative analgesia has not been fully understood and controlled, particularly craniotomy surgery. On the one hand, professional evaluation of postoperative pain for young children is difficult; on the other hand, the particularity of craniotomy adds (such as consciousness obstacle, sleepiness, et al) disturbance to the pain assessment in children. Although opioids administration is regarded as the first-line analgesic for post-craniotomy pain management, it may be associated with delayed awakening, respiratory depression, hypercarbia and it may interfere with the neurologic examination. For the avoidance of side-effects of systemic opioids, local anesthetics administered around the incision have been performed clinically. However, some studies revealed that the analgesic effect of local anesthetics was unsatisfactory due to its short pain relief duration, steroid as adjuvant can enhance postoperative analgesia and prolong postoperative analgesia time. As is reported that postoperative pain of craniotomy is mainly caused by skin incision and reflection of muscles, preventing the liberation of inflammatory mediators around the incision seems to be more effective than simply blocking nerve conduction. Thus, investigators suppose that pre-emptive scalp infiltration with steroid (Methylprednisolone) plus local anesthetic (ropivacaine) could relieve postoperative pain after craniotomy in children.

ELIGIBILITY:
Inclusion Criteria:

1. An elective craniotomy under general anesthesia;
2. American Society of Anesthesiologists (ASA) physical status of I or II;
3. Participates with an anticipated fully recovery within 2 hours postoperatively；
4. Informed consent by parent(s) and/or legal guardian.

Exclusion Criteria:

1. History of allergies to any of the study drugs;
2. Excessive alcohol or drug abuse, chronic opioids use (more than 2 weeks or 3 days per week for more than 1 month), or drugs with confirmed or suspected sedative or analgesic effects; receiving any painkiller within 24 h before surgery; children who received steroids；
3. Psychiatric disorders;
4. Uncontrolled epilepsy;
5. Chronic headache;
6. Peri-incisional infection;
7. Body mass index exceeded the 99th percentile for age;
8. Children who cannot use patient-controlled intravenous analgesia(PCIA) device;
9. Children who cannot understand an instruction of pain scales before surgery.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative fentanyl consumption within 24 hours postoperatively | Within 24 hours after the operation
  The PCIA device provides bolus (0.5µg/kg, 10min lock-out time) and the maximum dose will be limited as 2µg/kg per hour. If the patients feel inadequate analgesia after 5 times of fentanyl bolus, the bolus dose will be increased to 1 µg/kg and the maximum dose will be increased to 4 µg/kg per hour

SECONDARY OUTCOMES:
The number of participants who have no fentanyl consumption | Within 24 hours after the operation
  The number of participants who have not pushed the button of patient-controlled intravenous analgesia pump. Both of the initial dose and background infusion of the patient-controlled intravenous analgesia pump in this study will be set at 0. Participants will be advised to push the analgesic demand button if they feel pain.
The first time to press the patient-controlled intravenous analgesia button | Within 24 hours after the operation
  The first time that the participants press the patient-controlled intravenous analgesia button.
The total times that participants press patient-controlled intravenous analgesia button | Within 24 hours after the operation
  The total times that participants press patient-controlled intravenous analgesia button including effective presses and ineffective presses.
Numeric Rating Scale (NRS) | At 2 hours, 4 hours, 8 hours, 24 hours，48 hours, 72 hours, 1 week, 2 weeks, 1 month, 3 months, 6 months after surgery
  The NRS is a segmented numeric scale in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain. (0 indicates no pain, 10 indicates the most severe pain imaginable. Significant or moderate pain will be defined as NRS ≥4. Severe pain will be deﬁned as a pain score ≥7.
Pain control satisfaction score(PCSS) | At 24 hours，48 hours, 72 hours, 1 week, 2 weeks, 1 month, 3 months, 6 months after surgery
  PCSS (0 for unsatisfactory, and 10 for very satisfied) will be assessed patient satisfaction
length of stay (LOS) | At 24 hours，48 hours, 72 hours, 1 week, 2 weeks, 1 month, 3 months, 6 months after surgery
  LOS will be recorded as the number of nights spent in hospital after surgery.
The occurrence of postoperative nausea and vomiting | The duration of hospitalization after the operation
  Postoperative nausea and vomiting (PONV) was rated by participants as: 0, absent; 1, nausea not requiring treatment; 2, nausea requiring treatment; and 3, vomiting.
Ramsay Sedation Scale（RSS） | At 2 hours, 4 hours, 8 hours, 24 hours after surgery
  1: Anxious, agitated, restless; Ramsey 2: Cooperative, oriented, tranquil; Ramsey 3: Responsive to commands only If Asleep; Ramsey 4: Brisk response to light glabellar tap or loud auditory stimulus; Ramsey 5: Sluggish response to light glabellar tap or loud auditory stimulus; Ramsey 6: No response to light glabellar tap or loud auditory stimulus.Oversedation will be defined as a score of >2
The time to first water and oral intake request, scales of oral intake after operation | Within 24 hours after the operation
The occurrence of respiratory depression | Within 24 hours after the operation
  Respiratory depression is defined as persistent (more than 1 minutes) oxygen desaturation 90 percent or respiratory rate less than 8 breaths per minute, or oxygen desaturation less than 94 percent along with respiratory rate less than 10 breaths per minute requiring supplemental oxygen to maintain oxygen saturation more than 94 percent in the absence of clinically obvious upper airway obstruction.
Emergence delirium | Within 24 hours after the operation
  Emergence delirium will be assessed using the Pediatric Anesthesia Emergence Delirium (PAED) scale. (1) The child makes eye contact with the caregiver, (2) the child's actions are purposeful, (3) the child is aware of his/her surroundings, (4) the child is restless, and (5) the child is inconsolable. Items 1, 2, and 3 are reversed scored as follows: 4 not at all, 3 just a little, 2 quite a bit, 1 very much, 0 extremely. Items 4 and 5 are scored as follows: 0 not at all, 1 just a little, 2 quite a bit, 3 very much, 4 extremely. The scores of each item were summed to obtain a total PAED scale scores. Emergence agitation will be considered a total score of >12 at any time.
Heart rate | During the operation and at 2 hours, 4 hours, 8 hours, 24 hours after surgery
Mean arterial pressure | During the operation and at 2 hours, 4 hours, 8 hours, 24 hours after surgery
The total consumption of opioids during the operation | During procedure
The total consumption of anaesthetic during the operation | During procedure
Incisional related adverse events | Within 1 month after surgery
  Incisional related adverse events Including delayed incisional healing, incisional infection, intracranial infection, scar healing.
The occurrence of the Adverse events (AEs) and serious adverse events (SAEs) | Within 6 month after surgery
  An AE was defined as any untoward medical occurrence. An SAE included death, immediately life-threatening conditions, coma, in-patient hospitalisation or prolongation of existing hospitalisation.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao C, Jia Y, Jia Z, Xiao X, Luo F. Pre-emptive scalp infiltration with ropivacaine plus methylprednisolone versus ropivacaine alone for relief of postoperative pain after craniotomy in children (RP/MP vs RP): a study protocol for a randomised controlled trial. BMJ Open. 2019 Jun 22;9(6):e027864. doi: 10.1136/bmjopen-2018-027864. PMID 31230016